CLINICAL TRIAL: NCT01632878
Title: Omacor Plus Standard Therapies In Post MI Subjects Evaluation: The OPTIMISE Study
Brief Title: Omacor Plus Standard Therapies In Post Myocardial Infarction (MI) Subjects Evaluation: The OPTIMISE Observational Study
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: inVentiv Health Germany GmbH (Unknown); EBC - Evidence Based Communication (Unknown)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: P13-764
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2016-04

CONDITIONS: Myocardial Infarction (MI)
Keywords: Secondary prevention post MI
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post Myocardial Infarction: One single cohort of Index post Myocardial Infarction patients

SUMMARY:
The OPTIMISE study is a prospective, multi-center, multi-national, structured data collection initiative, first compiling data on the current treatment of post myocardial infarction patients (screening-log) and then, prospectively evaluating only those patients being prescribed Omacor as part of their standard secondary prevention treatment. The aim is to observe the Omacor cohort of patients for a period of 12 months, collecting long term observational data as clinical and patient-reported outcomes, especially, but not exclusively, recurrent non fatal Myocardial Infarction (MI), sudden death, or new Congestive Heart Failure (CHF). No predefined additional visits, medical tests, labs, procedures or interventions will be mandated. Only results from routinely performed tests, labs, procedures and/or interventions will be collected if available.

ELIGIBILITY:
Inclusion Criteria

* Male and female patients, from the screening-log, having been prescribed prior to their inclusion in the study Omega-3-fatty-acid ethyl esters (Omacor) as adjuvant treatment in secondary prevention after their myocardial infarction, in addition to standard therapy [e.g. statins, antiplatelet medicinal products, beta blockers, Angiotensine Converting Enzyme (ACE) inhibitors/Angiotensine II Receptor Blockers (ARBs), etc].

Exclusion Criteria

* Omega-3-fatty-acid ethyl esters (Omacor) approved contra-indication as per the labeling information in participating countries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 1531 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katinka Giezeman, Study Director — Mylan
Locations (1):
- Site Reference ID/Investigator# 81558, Plovdiv, Bulgaria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1531 patients were screened and the decision to treat patients with Omacor was made by the treating physician. 268 patients were not treated with Omacor according to the protocol. Only baseline characteristics were reported without any further follow-up for these patients.
Pre-assignment Details: 268 patients screened but not treated with Omacor on physician decision as per the protocol. Consequently 1263 entered in Omacor 1 year treatment assessment
Period: Screening
Arm/Group | Post Myocardial Infarction
Started | 1531
Completed | 1263
Not Completed | 268
Not completed — Physician Decision | 268
Period: Treatment
Arm/Group | Post Myocardial Infarction
Started | 1263
Completed | 1105
Not Completed | 158
Not completed — Lost to Follow-up | 41
Not completed — Withdrawal by Subject | 36
Not completed — Physician Decision | 34
Not completed — missing information | 4
Not completed — no information on study completion | 43

BASELINE CHARACTERISTICS:
Groups:
- Post Myocardial Infarction Omacor Group: Index post Myocardial Infarction patients screened and treated with Omacor as decided by physician
- Post Myocardial Infarction Non-Omacor Group: Index post Myocardial Infarction patients screened and not treated with Omacor as decided by physician
- Total: Total of all reporting groups
Arm/Group | Post Myocardial Infarction Omacor Group | Post Myocardial Infarction Non-Omacor Group | Total
Number analyzed (Participants) | 1263 | 268 | 1531
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.64) | 59.6 (11.37) | 59.2 (10.77)
Sex/Gender, Customized [Number; unit: participants]
  male | 948 | 203 | 1151
  female | 311 | 61 | 372
  unknown | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurrences of Cardio-vascular Events
Description: Such as: recurrent non fatal Myocardial Infarction (MI), sudden death, or new Congestive Heart Failure (CHF)
Time Frame: 12 months
Measure: Number; unit: events
Groups:
- Post Myocardial Infarction: Index post Myocardial Infarction patients (Omacor group)
Arm/Group | Post Myocardial Infarction
Number analyzed (Participants) | 1263
events
  Death | 4
  HF (Heart failure) | 3
  Recurrent, non-fatal myocardial infarction (RNFMI) | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Post Myocardial Infarction
Serious Adverse Events (participants affected / at risk) | 43/1263
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post Myocardial Infarction (N=1263)
Angina unstable (Cardiac disorders) | 9
Atrial fibrillation (Cardiac disorders) | 5
Coronary artery disease (Cardiac disorders) | 2
Pneumonia (Infections and infestations) | 2
Loss of consciousness (Nervous system disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 4
Atrioventricular block (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 2
Atrioventricular block first degree (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial fibrosis (Cardiac disorders) | 1
Postinfarction angina (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Aortic arteriosclerosis (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Adverse Events (non-serious) were not monitored in this observational study. This explains why 0/0 was reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No